CLINICAL TRIAL: NCT07069738
Title: Safety and Effectiveness of Left Bundle Branch Area Pacing Versus Conventional Cardiac Resynchronization Therapy in Heart Failure
Acronym: SYNCHRONICITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C2403
Record Dates: First submitted 2025-06-23; First posted 2025-07-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure - NYHA II - IV
Keywords: Heart Failure; Conduction System Pacing; Primary Prevention; Cardiac Resynchronization Therapy; Left Bundle Branch Area Pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CRT Cohort (Active Comparator): Participants will be randomized, implanted with a BSC CRT-D device using a Quadripolar lead, and device programmed to the respective cohort.
  Interventions: Device: CRT-D with a Quadripolar LV lead
- LBBA Cohort (Experimental): Participants will be randomized, implanted with a BSC CRT-D using the INGEVITY+ pace/sense lead implanted in the LBBA, and device programmed to the respective cohort.
  Interventions: Device: CRT-D with INGEVITY+ pace/sense lead

INTERVENTIONS:
Device: CRT-D with a Quadripolar LV lead — Participants randomized to this cohort will receive a BSC system: CRT-D, Right Atrial Lead (RA), Defibrillation Lead (RV), Quadripolar LV Lead.
  Arms: CRT Cohort
Device: CRT-D with INGEVITY+ pace/sense lead — Participants randomized to this cohort will receive a BSC system: CRT-D, Right Atrial Lead (RA), Defibrillation Lead (RV), INGEVITY+ pace/sense Lead (implanted in the LBBA)
  Arms: LBBA Cohort

SUMMARY:
This study will compare two different methods to pace the heart to treat heart failure including:

1. The current standard method of implanting a pacing lead in a vein on the surface of the left lower chamber of the heart (left ventricle) to deliver heart failure therapy. This method is called Cardiac Resynchronization Therapy (CRT).
2. The other method is using a lead implanted in the Left Bundle Branch Area (LBBA) of your heart. This method is called Left Bundle Branch Area Pacing or LBBAP. This lead is approved by the Food and Drug Administration (FDA) to be implanted in this area of the heart, but not to provide heart failure treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age 18 years or above, or of legal age to give informed consent specific to state and national law
2. Patient meets a guideline-based indication for a de novo CRT-D device
3. Primary prevention indication for ICD therapy
4. Ischemic or nonischemic cardiomyopathy with LVEF ≤ 35% within 6 months of enrollment (LVEF must be assessed after the subject has been on GDMT for a minimum of 3 months) using an appropriate method of assessment (i.e. Echo, MRI, etc)
5. NYHA class II-IV despite maximally tolerated guideline directed medical therapy (GDMT)* for at least 3 months

   *GDMT is defined as all four drug classes listed below for at least 3 months prior to enrollment unless the investigator provides justification (e.g., contraindicated, not tolerated or cost): Renin Angiotensin System Inhibitors (ACE, ARB, or ARNI) Evidence based betablockers (metoprolol succinate, carvedilol, bisoprolol) Mineralocorticoid antagonists SGLT2 Inhibitor medications
6. Sinus rhythm with left bundle branch block (LBBB) defined as a QRS ≥ 140 ms in men and ≥ 130 ms in women with a predominantly negative deflection (QS or rS in lead V1 and mid QRS notching or slurring in at least two of the following leads: 1, aVL, V1, V2, V5, V6) within 3 months of enrollment
7. Patient is willing to participate in LATITUDE™ NXT remote patient monitoring
8. Patient is willing and capable of providing informed consent and participating in all testing associated with this investigation at an approved study site and at the protocol defined intervals (Note: Use of a legally authorized representative (LAR) is not allowed)
9. Patient plans to remain geographically stable (not permanently moving to another location) and can commit to all study participation requirements (procedure, follow-up visits and testing requirements)

Exclusion Criteria:

1. Persistent or permanent atrial fibrillation (AF) within 3 months prior to enrollment and documented in the medical record
2. Frequent premature ventricular contractions (PVCs), atrial arrhythmias, and/or other causes of expected percentage of cardiac physiologic pacing (CPP) delivery below 95% at the time of enrollment
3. Non-LBBB conduction abnormalities (including right bundle branch block (RBB) or intraventricular conduction delay (IVCD)) within 3 months prior to enrollment
4. Complete, second degree or high degree atrioventricular (AV) block, that requires pacing at the time of enrollment
5. Current or prior pacemaker, ICD or CRT implant (Also includes non-transvenous ICD technology and leadless pacemakers)
6. Prior or planned mechanical or bioprosthetic tricuspid valve replacement
7. Currently receiving or previously received positive inotrope therapy within 3 months prior to enrollment
8. Unstable angina, acute myocardial infarction, coronary artery bypass grafting, or percutaneous coronary intervention within 3 months prior to enrollment
9. History of heart transplantation or left ventricular assist device (LVAD) implantation
10. Less than 1 year of life expectancy at the time of enrollment
11. Anticipated heart transplantation or LVAD implantation within 1 year of enrollment
12. History of ventricular septal defect (VSD)
13. Complex congenital heart disease
14. Documented diagnosis of cardiac amyloidosis
15. Known occlusion or other reason limiting central venous access for transvenous leads
16. Women of childbearing potential who are, or plan to become, pregnant during the course of the study (assessment per investigator's discretion)
17. Patient currently requiring dialysis
18. Patient with known or suspected sensitivity to Dexamethasone Acetate (DXA)
19. Patient with contrast dye allergy or unwilling/able to undergo pre-treatment with steroids and/or diphenhydramine
20. Inability or refusal to comply with the follow-up schedule including subject living at such a distance from the investigational site that attending follow-up visits would be unusually difficult or burdensome
21. Patient is enrolled in any other concurrent study. Co-enrollment into other studies such as observational studies/registries needs prior written approval by BSC. Local mandatory governmental registries are accepted for co-enrollment without approval by BSC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Composite of reduction in all-cause mortality, heart transplant, left ventricular assist device, heart failure events, ventricular tachycardia/ventricular fibrillation requiring device therapy or external defibrillation/cardioversion. | Through study completion, up to maximum of 5 years
  The primary effectiveness endpoint is a composite of reduction in all-cause mortality, heart transplant, left ventricular assist device (LVAD), time to first heart failure (HF) events, time to first ventricular tachycardia (VT) / ventricular fibrillation (VF) requiring device therapy or external defibrillation/cardioversion.
System-related complication-free rate | 12 months
  The primary safety endpoint is System-related complication-free rate of LBBAP at 12 months. This will be a single-arm analysis of the LBBAP group compared to a performance goal

SECONDARY OUTCOMES:
Win ratio composite assessment | Through study completion, up to a maximum of 5 years
  Win Ratio Ranking: 1) Death 2) Heart Transplant/LVAD 3) Number of Heart Failure (HF) events (includes in-patient, out-patient and HF re-admission 4) Number of VT/VF episodes requiring device therapy or external defibrillation/cardioversion (one episode per 24 hours 5) Change in MLHFQ (Minnesota Living with Heart Failure Questionnaire) quality of life
Composite of reduction in all-cause mortality, heart transplant, left ventricular assist device, heart failure events, ventricular tachycardia/ ventricular fibrillation requiring device therapy or external defibrillation/cardioversion. | Through study completion, up to a maximum of 5 years
  The primary effectiveness endpoint is a composite of reduction in all-cause mortality, heart transplant, left ventricular assist device (LVAD), time to first heart failure (HF) events, time to first ventricular tachycardia (VT) / ventricular fibrillation (VF) requiring device therapy or external defibrillation/cardioversion.
System-related complication-free rate between randomized arms | 12 months
  System-related complication-free rate of LBBAP at 12 months. This will compare the two randomized arms.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Alta Bates Summit Medical Center, Oakland, California
  - Cardiology Associates Medical Group, Inc., Ventura, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Centracare Heart and Vascular Center, Saint Cloud, Minnesota
  - New York Hospital Queens, Flushing, New York
  - Weill Cornell Medical University, New York, New York
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Christus Trinity Mother Frances Health System, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No